CLINICAL TRIAL: NCT03910686
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation and Cognitive Behavioral Therapy on Alcohol Dependence
Acronym: TAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ying Peng, Professor, Director of Department of Neurology, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-12-TMSCBT
Record Dates: First submitted 2019-04-03; First posted 2019-04-10 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Dependence, transcranial magnetic stimulation, cognitive behavioral therapy
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Magnetic Stimulation; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Regular treatment (symptomatic treatment) with blank TMS (Placebo Comparator): Regular treatment (symptomatic treatment) with blank transcranial magnetic stimulation
  Interventions: Combination Product: Transcranial magnetic stimulation and cognitive behavioral therapy
- Regular treatment (RT) with blank TMS and CBT (Active Comparator): Regular treatment (symptomatic treatment) with blank transcranial magnetic stimulation and cognitive behavioral therapy
  Interventions: Combination Product: Transcranial magnetic stimulation and cognitive behavioral therapy
- RT with right DLPFC hf-rTMS (Active Comparator): Regular treatment with right dorsolateral prefrontal cortex (DLPFC) high frequency repetitive transcranial magnetic stimulation (hf-rTMS)
  Interventions: Combination Product: Transcranial magnetic stimulation and cognitive behavioral therapy
- RT with right DLPFC hf-rTMS and CBT (Active Comparator): Regular treatment with right DLPFC high frequency repetitive transcranial magnetic stimulation (hf-rTMS) and cognitive behavioral therapy (CBT)
  Interventions: Combination Product: Transcranial magnetic stimulation and cognitive behavioral therapy
- RT with left DLPFC hf-rTMS (Active Comparator): Regular treatment with left DLPFC high frequency repetitive transcranial magnetic stimulation (hf-rTMS)
  Interventions: Combination Product: Transcranial magnetic stimulation and cognitive behavioral therapy
- RT with left DLPFC hf-rTMS and CBT (Active Comparator): Regular treatment with left DLPFC high frequency repetitive transcranial magnetic stimulation (hf-rTMS) and cognitive behavioral therapy (CBT)
  Interventions: Combination Product: Transcranial magnetic stimulation and cognitive behavioral therapy

INTERVENTIONS:
Combination Product: Transcranial magnetic stimulation and cognitive behavioral therapy — Transcranial magnetic stimulation on different side with/without cognitive behavioral therapy

SUMMARY:
Alcohol dependence is one of most common substance dependence, which brings great burden on health worldwide. Alcohol dependence may lead to many serious diseases or consequences including cancer, cardiovascular diseases and accidents. Once alcohol dependence is developed, it will be difficult to recover and easy to relapse. Although many efforts had been made in the treatment of alcohol dependence, the annual recurrence of alcohol dependence with traditional therapies was over 45%. Repetitive transcranial magnetic stimulation (rTMS) on the dorsolateral prefrontal cortex (DLPFC) or cognitive behavioral therapy (CBT) each alone was reported to have some effect on preventing from relapse of alcohol dependence. In order to test whether combined therapy of high frequency rTMS (hf-rTMS) with CBT is better for preventing from relapse of alcohol dependence, we recruit patients with alcohol dependence to participate this study. The study is a factorial designed and the patients will be assigned into one of the following six groups randomly: (1) regular treatment (symptomatic treatment) with blank TMS; (2) regular treatment (RT) with blank TMS and CBT; (3) RT with right DLPFC hf-rTMS; (4) RT with right DLPFC hf-rTMS and CBT; (5) RT with left DLPFC hf-rTMS; (6) RT with left DLPFC hf-rTMS and CBT. TMS was given 5 days per week for total 2 weeks using uniform scheme (5 seconds of 10Hz stimulation per train, 30 trains per day with inter-train interval of 20 seconds). CBT will be given once per week for total 8 weeks. The patients will be followed up for 6 months. Recurrence of alcohol dependence, duration of abstention, alcohol intake, craving for alcohol and other cognitive psychological assessments will be recorded and compared among the 6 treatment groups and the efficacy of combined therapy of rTMS with CBT will be evaluated in our study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis as alcohol dependence according to DSM-IV criteria
* No definite history of neurological diseases and psychological problems
* Volunteer to participate the study, cooperate to be followed up

Exclusion Criteria:

* Acute withdrawal state and CIWA score > 9
* With other neurological diseases and psychological problems
* With ever brain trauma and damage
* With other psychological medications or other substance dependence
* With other contraindications to have transcranial magnetic stimulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The rate of relapse of alcohol dependence after discharge from hospital | 1 month
  Recurrence of alcohol dependence
The rate of relapse of alcohol dependence after discharge from hospital | 2 month
The rate of relapse of alcohol dependence after discharge from hospital | 3 month
The rate of relapse of alcohol dependence after discharge from hospital | 6 month

SECONDARY OUTCOMES:
Duration of abstinence | 6 months
  The total time or period without any intake of alcohol during follow ups
Alcohol intake | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Diaries of alcohol intake in different time of the follow ups
Craving for alcohol | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Craving assessment for alcohol by Obsessive Compulsive Drinking Scale (OCDS) ranging from 0 to 40. Higher score of OCDS indicates more desire for alcohol.
Craving for alcohol | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Craving assessment by Visual Analogue Scale (VAS) for alcohol desire ranging from 0 to 10. Higher score indicates more desire for alcohol.
Cognitive assessment | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Cognitive assessment by Montreal Cognitive Assessment (MoCA) ranging from 0 to 30. Lower score indicates worse cognitive function.
Psychological assessment - Anxiety | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Psychological assessment by Generalized Anxiety Disorder-7 (GAD-7) ranging from 0 to 21. Higher score indicates more severer anxiety.
Psychological assessment - Depression | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Psychological assessment by Patient Health Questionnaire-9 (PHQ-9) ranging from 0 to 27. Higher score indicates more severer depression.
Psychological assessment - Sleep | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Psychological assessment by Pittsburgh Sleep Quality Index (PSQI) ranging from 0 to 21. Higher score indicates worse sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips MR, Zhang J, Shi Q, Song Z, Ding Z, Pang S, Li X, Zhang Y, Wang Z. Prevalence, treatment, and associated disability of mental disorders in four provinces in China during 2001-05: an epidemiological survey. Lancet. 2009 Jun 13;373(9680):2041-53. doi: 10.1016/S0140-6736(09)60660-7. PMID 19524780
- [Background] Tang YL, Hao W, Leggio L. Treatments for alcohol-related disorders in China: a developing story. Alcohol Alcohol. 2012 Sep-Oct;47(5):563-70. doi: 10.1093/alcalc/ags066. Epub 2012 Jun 7. PMID 22683652
- [Background] Mishra BR, Nizamie SH, Das B, Praharaj SK. Efficacy of repetitive transcranial magnetic stimulation in alcohol dependence: a sham-controlled study. Addiction. 2010 Jan;105(1):49-55. doi: 10.1111/j.1360-0443.2009.02777.x. PMID 20078462
- [Background] Herremans SC, Vanderhasselt MA, De Raedt R, Baeken C. Reduced intra-individual reaction time variability during a Go-NoGo task in detoxified alcohol-dependent patients after one right-sided dorsolateral prefrontal HF-rTMS session. Alcohol Alcohol. 2013 Sep-Oct;48(5):552-7. doi: 10.1093/alcalc/agt054. Epub 2013 May 24. PMID 23709633
- [Background] Mishra BR, Praharaj SK, Katshu MZ, Sarkar S, Nizamie SH. Comparison of anticraving efficacy of right and left repetitive transcranial magnetic stimulation in alcohol dependence: a randomized double-blind study. J Neuropsychiatry Clin Neurosci. 2015 Winter;27(1):e54-9. doi: 10.1176/appi.neuropsych.13010013. PMID 25255169
- [Background] Herremans SC, De Raedt R, Van Schuerbeek P, Marinazzo D, Matthys F, De Mey J, Baeken C. Accelerated HF-rTMS Protocol has a Rate-Dependent Effect on dACC Activation in Alcohol-Dependent Patients: An Open-Label Feasibility Study. Alcohol Clin Exp Res. 2016 Jan;40(1):196-205. doi: 10.1111/acer.12937. PMID 26727534
- [Background] Sundstrom C, Kraepelien M, Eek N, Fahlke C, Kaldo V, Berman AH. High-intensity therapist-guided internet-based cognitive behavior therapy for alcohol use disorder: a pilot study. BMC Psychiatry. 2017 May 26;17(1):197. doi: 10.1186/s12888-017-1355-6. PMID 28549424